CLINICAL TRIAL: NCT07398612
Title: Clinical Study on the Safety and Efficacy of Human Adipose-Derived Stem Cell Exosomes in the Treatment of Acute Ischemic Stroke
Brief Title: Safety and Efficacy of Human Adipose-Derived Stem Cell Exosomes in Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai 10th People's Hospital (Other); First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yuncheng Wu, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT-ATMP-2025011
Record Dates: First submitted 2025-12-30; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; human adipose-derived stem cell; exosome; NIHSS; mRS
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This is an interventional clinical trial model that sequentially combines two distinct designs within a single protocol:
  An open-label, sequential cohort, single-ascending dose (SAD) design for initial dose-finding and safety profiling. It uses a modified "3+3" type logic (4 subjects per cohort) with predefined safety stopping rules to guide dose escalation between cohorts.
  A randomized, double-blind, parallel-group, multiple-ascending dose (MAD) design with placebo control for preliminary efficacy evaluation and further safety assessment. It features two sequentially enrolled dose cohorts (low and high), each with an internal 2:1 randomization (active:placebo). Progression from the low-dose to the high-dose cohort is contingent upon a safety review, making it a sequential cohort expansion within the randomized phase.
  This hybrid model is typical for early-phase trials of novel biological therapies, aiming to efficiently establish a safe dose range (SAD) before exploring preliminary
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a double-blind design. The following parties are masked (blinded):
  Subjects: Participants will not know whether they are receiving ADSC-exo or placebo (saline).
  Investigators and Site Staff: All personnel directly involved in treating subjects, evaluating clinical outcomes (including efficacy scale assessments), and managing subject care during the trial will be blinded to treatment assignment. This includes the Principal Investigator, sub-investigators, and study nurses.
  Sponsor's Clinical Team: Personnel from the sponsor involved in the day-to-day monitoring and clinical operations of the trial will remain blinded.
  To maintain the blind, the active drug (ADSC-exo solution) and the placebo (saline) are prepared to be identical in appearance, packaging, and labeling. An interactive web response system (IWRS) will manage randomization and drug kit assignment. The sponsor will designate a limited number of unblinded personnel (e.g., an unblinded statistician respon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Single Ascending Dose Study Cohort 1 (Experimental): This is an open-label, single-dose cohort in the dose-escalation phase (Part 1). Four (4) subjects with acute ischemic stroke will receive a single dose of Human Adipose-Derived Stem Cell Exosomes (ADSC-exo) Nasal Spray at a concentration of 2×10^9 particles per mL (total volume 1 mL), administered intranasally once.
  Interventions: Biological: Human Adipose-Derived Stem Cell Exosomes
- Single Ascending Dose Study Cohort 2 (Experimental): This is an open-label, single-dose cohort in the dose-escalation phase (Part 1). Four (4) subjects with acute ischemic stroke will receive a single dose of Human Adipose-Derived Stem Cell Exosomes (ADSC-exo) Nasal Spray at a concentration of 4×10^9 particles per mL (total volume 1 mL), administered intranasally once.
  Interventions: Biological: Human Adipose-Derived Stem Cell Exosomes
- Single Ascending Dose Study Cohort 3 (Experimental): This is an open-label, single-dose cohort in the dose-escalation phase (Part 1). Four (4) subjects with acute ischemic stroke will receive a single dose of Human Adipose-Derived Stem Cell Exosomes (ADSC-exo) Nasal Spray at a concentration of 8×10^9 particles per mL (total volume 1 mL), administered intranasally once.
  Interventions: Biological: Human Adipose-Derived Stem Cell Exosomes
- Multiple Dose Study Low-Dose ADSC-exo (X) (Experimental): This is a double-blind, multiple-dose treatment arm in the dose-expansion phase (Part 2). Sixteen (16) subjects with acute ischemic stroke will receive Human Adipose-Derived Stem Cell Exosomes (ADSC-exo) Nasal Spray at a low concentration (designated as X ×10^9 particles per mL, to be determined based on SAD results), administered intranasally once daily (QD) for 14 consecutive days. This is administered in addition to standard of care (SOC). This arm is compared to a placebo control arm within the same low-dose group.
  Interventions: Biological: Human Adipose-Derived Stem Cell Exosomes
- Multiple Dose Study Low-Dose Placebo (Placebo Comparator): This is a double-blind, multiple-dose control arm in the dose-expansion phase (Part 2). Eight (8) subjects with acute ischemic stroke will receive a matching Placebo Nasal Spray (0.9% physiological saline), administered intranasally once daily (QD) for 14 consecutive days. This is administered in addition to standard of care (SOC). This arm serves as the comparator for the active low-dose ADSC-exo arm.
  Interventions: Other: Placebo
- Multiple Dose Study High-Dose ADSC-exo (Y) (Experimental): This is a double-blind, multiple-dose treatment arm in the dose-expansion phase (Part 2). Sixteen (16) subjects with acute ischemic stroke will receive Human Adipose-Derived Stem Cell Exosomes (ADSC-exo) Nasal Spray at a high concentration (designated as Y ×10^9 particles per mL, to be determined based on SAD results), administered intranasally once daily (QD) for 14 consecutive days. This is administered in addition to standard of care (SOC). This arm is compared to a placebo control arm within the same high-dose group. Enrollment into this high-dose group is contingent upon a safety review of the low-dose group.
  Interventions: Biological: Human Adipose-Derived Stem Cell Exosomes
- Multiple Dose Study High-Dose Placebo (Placebo Comparator): This is a double-blind, multiple-dose control arm in the dose-expansion phase (Part 2). Eight (8) subjects with acute ischemic stroke will receive a matching Placebo Nasal Spray (0.9% physiological saline), administered intranasally once daily (QD) for 14 consecutive days. This is administered in addition to standard of care (SOC). This arm serves as the comparator for the active high-dose ADSC-exo arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Human Adipose-Derived Stem Cell Exosomes — This intervention involves the use of allogeneic Human Adipose-Derived Stem Cell Exosomes (ADSC-exo), provided as a sterile nasal spray (STX11102).
  Arms: Multiple Dose Study High-Dose ADSC-exo (Y); Multiple Dose Study Low-Dose ADSC-exo (X); Single Ascending Dose Study Cohort 1; Single Ascending Dose Study Cohort 2; Single Ascending Dose Study Cohort 3
Other: Placebo — This intervention serves as the placebo control. It is a sterile 0.9% sodium chloride (normal saline) solution formulated as a nasal spray
  Arms: Multiple Dose Study High-Dose Placebo; Multiple Dose Study Low-Dose Placebo

SUMMARY:
This is a Phase I/II, randomized, double-blind, placebo-controlled, single/multiple ascending dose clinical study (Investigator-Initiated Trial, IIT) evaluating the safety and efficacy of Human Adipose-Derived Stem Cell Exosomes (ADSC-exo, STX11102 Nasal Spray) in treating acute ischemic stroke (AIS). The study consists of two sequential parts: a Single-Ascending Dose (SAD) study and a Multiple-Ascending Dose (MAD) study.

The SAD part will enroll 12 subjects with mild stroke (NIHSS 1-4). They will be sequentially enrolled into three dose cohorts (4 subjects each: 2×10⁹, 4×10⁹, and 8×10⁹ particles/mL) to receive a single nasal spray dose alongside standard care, with safety monitoring for 14 days. Dose escalation is contingent upon the safety review of the preceding cohort.

Upon confirming safety, the study proceeds to the MAD part, which will enroll 48 subjects with moderate stroke (NIHSS 5-12). They will be randomized into two dose groups (Low and High Dose), each containing an active treatment arm and a placebo arm (saline) in a 2:1 ratio (16 active:8 placebo per group). Subjects will self-administer the nasal spray daily for 14 days, with follow-up until Day 90. The primary objective is to evaluate safety, with secondary objectives assessing efficacy via neurological function scales (NIHSS, mRS, BI) and infarct volume change on MRI.

DETAILED DESCRIPTION:
This clinical trial is designed to investigate the novel therapeutic agent Human Adipose-Derived Stem Cell Exosomes (ADSC-exo, STX11102) delivered via nasal spray for patients with acute ischemic stroke (AIS). The rationale is based on promising preclinical data demonstrating that intranasally administered ADSC-exo can cross the blood-brain barrier, modulate neuroinflammation, reduce infarct volume, and promote functional recovery in animal stroke models.

Study Design and Phases:

The trial employs a two-part, early-phase exploratory design integrating dose-finding and preliminary efficacy assessment.

Part 1: Single-Ascending Dose (SAD) Study: This is an open-label, dose-escalation phase to assess initial safety and tolerability. Twelve subjects with mild AIS (NIHSS 1-4, onset within 72 hours) will be enrolled at a single center. Three dose levels will be tested sequentially: Dose Cohort 1 (2×10⁹ particles/mL), Cohort 2 (4×10⁹ particles/mL), and Cohort 3 (8×10⁹ particles/mL), with 4 subjects per cohort. All subjects will receive a single dose of ADSC-exo nasal spray plus standard care. Escalation to the next higher dose cohort requires completion of the 14-day safety observation for all subjects in the current cohort and a formal safety review by the Principal Investigator (PI) and the sponsor. Escalation is permitted only if the number of subjects experiencing Grade ≥3 adverse events (AEs) considered related to the study drug is ≤50% (i.e., ≤2 subjects) within the completed cohort.

Part 2: Multiple-Ascending Dose (MAD) Study: This is a randomized, double-blind, placebo-controlled, dose-expansion phase to further evaluate safety and explore efficacy. Forty-eight subjects with moderate AIS (NIHSS 5-12, onset within 72 hours) will be enrolled across approximately five centers. Entry into this part requires a favorable safety review of all data from the SAD part. Subjects will be randomized into two sequential dose groups (Low Dose and High Dose). The specific doses (X and Y ×10⁹ particles/mL) for the MAD part will be determined based on SAD results. Each dose group consists of 24 subjects randomized in a 2:1 ratio to receive either ADSC-exo nasal spray (n=16) or matching placebo (saline, n=8) daily for 14 days, in addition to standard care. The Low Dose group must complete enrollment and 14-day safety follow-up before the High Dose group begins enrollment, applying the same safety criteria (≤50% of subjects with related Grade ≥3 AEs) for progression.

Study Population: Key inclusion criteria: age 18-80, anterior circulation ischemic stroke, pre-stroke mRS ≤1. Key exclusion criteria: severe stroke (NIHSS >12), lacunar/brainstem/cerebellar infarct, need for endovascular intervention, intracranial hemorrhage, malignancy, immunodeficiency, significant hepatic/renal impairment, active severe infection, and positive serology for HIV, HBV (with positive DNA), HCV, or syphilis.

Endpoints:

Primary Safety Endpoints: Incidence, severity, and causality of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs); changes in nasal mucosa, pulmonary function, and immunoglobulins.

Secondary Efficacy Endpoints:

SAD: Change from baseline in NIHSS, mRS, and Barthel Index (BI) at Day 14.

MAD: Change in NIHSS at Day 14; change in mRS and BI at Days 7, 14, 30, and 90; change in cerebral infarct lesion volume on MRI at Day 90.

Exploratory Endpoints (MAD): Changes in inflammatory cytokines (IL-2, IL-6, IL-12, IL-1β, TNF-α, IFN-γ).

Study Procedures: The schedule includes a 7-day screening period, treatment period (1 day for SAD, 14 days for MAD), and a follow-up period (14 days for SAD, 76 days for MAD). Assessments include neurological scales (NIHSS, mRS, BI), laboratory tests, vital signs, ECGs, MRI, and pulmonary function tests.

Statistical Analysis: This is an exploratory study with a sample size based on clinical practice. Safety will be analyzed in the Safety Set (SS). Efficacy will be analyzed descriptively for the SAD part. For the MAD part, efficacy will be analyzed in the Full Analysis Set (FAS) and Intent-to-Treat (ITT) set using appropriate statistical models (e.g., ANCOVA for continuous endpoints, Cochran-Mantel-Haenszel test for

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, male or female
2. Patients with acute ischemic stroke within 72 hours of symptom onset
3. Internal carotid artery system stroke
4. For the single-dose study: mild stroke patients (NIHSS score 1-4, inclusive of 1 and 4)
5. For the multiple-dose study: moderate stroke patients (NIHSS score 5-12, inclusive of 5 and 12)
6. Pre-stroke mRS score ≤ 1
7. Subjects or their guardians voluntarily sign the informed consent form

Exclusion Criteria:

1. Moderate or severe stroke (NIHSS score > 12).
2. Lacunar infarction, brainstem or cerebellar infarction (confirmed by DWI-MRI).
3. Requirement for endovascular interventional treatment for the current episode.
4. Intracranial hemorrhagic diseases (including parenchymal, intraventricular, subarachnoid hemorrhage, etc.).
5. Patients with malignant tumors.
6. Patients with severe traumatic brain injury.
7. Patients with primary or secondary immunodeficiency diseases or requiring immunosuppressant medication.
8. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding 3 times the upper limit of normal.
9. Chronic kidney disease or current serum creatinine exceeding 1.5 times the upper limit of normal or estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m².
10. Presence of severe infection or fever; patients with severe respiratory diseases.
11. Positive for hepatitis B virus surface antigen (HBsAg); or positive for hepatitis B core antibody (HBcAb) with positive HBV-DNA; or positive for hepatitis C virus antibody (HCVAb), Treponema pallidum antibody (TPAb/RPR), or human immunodeficiency virus antibody (HIV).
12. Patients who are pregnant or lactating at screening, or wish to become pregnant during the study period. Patients allergic to the product
13. Patients allergic to the product or with severe allergic constitution.
14. Patients deemed unsuitable for participation by the investigator, or for whom participation may pose a greater risk.
15. Patients who have participated in another clinical trial within the past 3 months.
16. Patients with prior use of exosomes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke. | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs): The incidence, severity (graded per CTCAE v5.0), and the investigator-assessed causality (relationship to the study drug) of all AEs and SAEs occurring during the treatment and follow-up period.
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke. | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Specific Safety Assessments:
  Nasal Mucosa: Changes from baseline based on physical examination of the nasal cavity.
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke. | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Specific Safety Assessments: pulmonary function: Changes in FVC versus baseline
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Specific Safety Assessments: pulmonary function: Changes in FEV versus baseline
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Specific Safety Assessments: pulmonary function: Changes in PEF versus baseline
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke. | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Immunoglobulins: Changes from baseline in serum levels of IgA.
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke. | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Immunoglobulins: Changes from baseline in serum levels of IgE
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Immunoglobulins: Changes from baseline in serum levels of IgM.
Safety and Tolerability of ADSC-exo Nasal Spray in Acute Ischemic Stroke | For Single-Dose Study: From first dose on Day 1 through the end of safety follow-up at Day 14. For Multiple-Dose Study: From first dose on Day 1 through the end of safety follow-up, which extends up to 14 days after the last dose on Day 14.
  Immunoglobulins: Changes from baseline in serum levels of IgG.

SECONDARY OUTCOMES:
Change in Neurological Function (For Single-Dose Study) | Baseline (Day 1, pre-dose) to Day 14 post-dose.
  This outcome measures the effect of a single dose of ADSC-exo on neurological recovery in patients with mild acute ischemic stroke (NIHSS 1-4). The change from baseline will be assessed using three validated clinical scales at Day 14 post-dose: the National Institutes of Health Stroke Scale (NIHSS) for stroke severity.The scoring range is 0-42 points, with higher scores indicating more severe nerve damage.
Change in NIHSS Score after 14-Day Treatment (For Multiple-Dose Study) | Baseline (Day 1, pre-dose) to Day 14 (end of treatment).
  This outcome measures the change in stroke severity after 14 days of multiple-dose treatment with ADSC-exo in patients with moderate acute ischemic stroke (NIHSS 5-12). The National Institutes of Health Stroke Scale (NIHSS) score will be compared from baseline (Day 1) to the end of the 14-day treatment period (Day 14). A decrease in NIHSS score indicates an improvement in neurological deficit.The scoring range is 0-42 points, with higher scores indicating more severe nerve damage.
Change in Disability & Daily Function (For Multiple-Dose Study) | Baseline (Day 1, pre-dose) to Day 7, Day 14, Day 30, and Day 90.
  This outcome measures the sustained effect of multiple-dose ADSC-exo treatment on global disability and daily living function over time. The change from baseline will be assessed using the modified Rankin Scale (mRS) for disability and the Barthel Index (BI) for activities of daily living at multiple timepoints: Day 7, Day 14, Day 30, and Day 90. Lower mRS scores(The scoring range is 0-6 points) and higher BI scores(The scoring range is 0-100 points) indicate better functional outcomes.
Change in Cerebral Infarct Volume on MRI (For Multiple-Dose Study) | Baseline MRI (within screening period, Day -7 to -1) to Day 90 MRI.
  This outcome is an imaging-based measure of treatment efficacy. It assesses the change in the volume of the cerebral infarct lesion from baseline (pre-treatment) to 90 days after the start of treatment (Day 90) using Magnetic Resonance Imaging (MRI). A reduction in infarct volume is hypothesized to correlate with neurological recovery and is a key structural endpoint.
Change in Neurological Function (For Single-Dose Study) | Baseline (Day 1, pre-dose) to Day 14 post-dose.
  This outcome measures the effect of a single dose of ADSC-exo on neurological recovery in patients with mild acute ischemic stroke (NIHSS 1-4). The change from baseline will be assessed using the validated clinical scales at Day 14 post-dose: the modified Rankin Scale (mRS) for global disability.The scoring range is 0-6 points, with higher scores indicating more severe nerve damage.
Change in Neurological Function (For Single-Dose Study) | Baseline (Day 1, pre-dose) to Day 14 post-dose.
  This outcome measures the effect of a single dose of ADSC-exo on neurological recovery in patients with mild acute ischemic stroke (NIHSS 1-4). The change from baseline will be assessed using the validated clinical scales at Day 14 post-dose:the Barthel Index (BI) for activities of daily living. The scoring range is 0-100 points, with higher BI scores indicate better functional outcomes.

IPD SHARING:
Plan to Share IPD: Yes
This study will share de-identified individual participant data (IPD) that underlies the results reported in the primary and secondary outcome publications. This will include baseline characteristics (e.g., age, sex, NIHSS score at entry, pre-stroke mRS), treatment assignment (dose group), and outcome data for all primary and secondary endpoints. Specifically, shared data will encompass safety endpoints (all recorded Treatment-Emergent Adverse Events, Serious Adverse Events, and changes in nasal mucosa, pulmonary function, and immunoglobulins) and efficacy endpoints (serial assessments of NIHSS, mRS, Barthel Index scores, and cerebral infarct volume change on MRI at Day 90 for the MAD part). All shared data will be fully anonymized to protect participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified IPD, study protocol, SAP, and ICF will become available 12 months after the publication of the primary study results (anticipated around September 2029, based on the Study Completion date of August 31, 2028). The data will be accessible for a period of 5 years thereafter (anticipated until September 2034). Requests can be submitted during this 5-year window.
Access Criteria: Access will be granted to qualified researchers from accredited scientific or medical institutions for the purpose of conducting analyses to achieve pre-specified research goals in the approved proposal. Examples include independent validation of results, meta-analysis, or exploration of novel scientific questions. Requestors must submit a methodologically sound research proposal through the designated access portal.
URL: https://clinicaltrials.gov/

REFERENCES:
- [Background] Xie X, Song Q, Dai C, Cui S, Tang R, Li S, Chang J, Li P, Wang J, Li J, Gao C, Chen H, Chen S, Ren R, Gao X, Wang G. Clinical safety and efficacy of allogenic human adipose mesenchymal stromal cells-derived exosomes in patients with mild to moderate Alzheimer's disease: a phase I/II clinical trial. Gen Psychiatr. 2023 Oct 11;36(5):e101143. doi: 10.1136/gpsych-2023-101143. eCollection 2023. PMID 37859748
- [Background] Li Y, Tang Y, Yang GY. Therapeutic application of exosomes in ischaemic stroke. Stroke Vasc Neurol. 2021 Sep;6(3):483-495. doi: 10.1136/svn-2020-000419. Epub 2021 Jan 11. PMID 33431513
- [Background] Sonoda T, Matsuzaki J, Yamamoto Y, Sakurai T, Aoki Y, Takizawa S, Niida S, Ochiya T. Serum MicroRNA-Based Risk Prediction for Stroke. Stroke. 2019 Jun;50(6):1510-1518. doi: 10.1161/STROKEAHA.118.023648. Epub 2019 Apr 15. PMID 31136284
- [Background] Dehghani L, Khojasteh A, Soleimani M, Oraee-Yazdani S, Keshel SH, Saadatnia M, Saboori M, Zali A, Hashemi SM, Soleimani R. Safety of Intraparenchymal Injection of Allogenic Placenta Mesenchymal Stem Cells Derived Exosome in Patients Undergoing Decompressive Craniectomy Following Malignant Middle Cerebral Artery Infarct, A Pilot Randomized Clinical Trial. Int J Prev Med. 2022 Jan 19;13:7. doi: 10.4103/ijpvm.ijpvm_441_21. eCollection 2022. PMID 35281985
- [Background] Yang Y, Cai Y, Zhang Y, Liu J, Xu Z. Exosomes Secreted by Adipose-Derived Stem Cells Contribute to Angiogenesis of Brain Microvascular Endothelial Cells Following Oxygen-Glucose Deprivation In Vitro Through MicroRNA-181b/TRPM7 Axis. J Mol Neurosci. 2018 May;65(1):74-83. doi: 10.1007/s12031-018-1071-9. Epub 2018 Apr 29. PMID 29705934
- [Background] Yang J, Zhang X, Chen X, Wang L, Yang G. Exosome Mediated Delivery of miR-124 Promotes Neurogenesis after Ischemia. Mol Ther Nucleic Acids. 2017 Jun 16;7:278-287. doi: 10.1016/j.omtn.2017.04.010. Epub 2017 Apr 13. PMID 28624203
- [Background] Xin H, Katakowski M, Wang F, Qian JY, Liu XS, Ali MM, Buller B, Zhang ZG, Chopp M. MicroRNA cluster miR-17-92 Cluster in Exosomes Enhance Neuroplasticity and Functional Recovery After Stroke in Rats. Stroke. 2017 Mar;48(3):747-753. doi: 10.1161/STROKEAHA.116.015204. PMID 28232590
- [Background] Altmann P, Mildner M, Haider T, Traxler D, Beer L, Ristl R, Golabi B, Gabriel C, Leutmezer F, Ankersmit HJ. Secretomes of apoptotic mononuclear cells ameliorate neurological damage in rats with focal ischemia. F1000Res. 2014 Jun 19;3:131. doi: 10.12688/f1000research.4219.2. eCollection 2014. PMID 25383184
- [Background] Hayon Y, Dashevsky O, Shai E, Brill A, Varon D, Leker RR. Platelet microparticles induce angiogenesis and neurogenesis after cerebral ischemia. Curr Neurovasc Res. 2012 Aug;9(3):185-92. doi: 10.2174/156720212801619018. PMID 22621230
- [Background] Chen KH, Chen CH, Wallace CG, Yuen CM, Kao GS, Chen YL, Shao PL, Chen YL, Chai HT, Lin KC, Liu CF, Chang HW, Lee MS, Yip HK. Intravenous administration of xenogenic adipose-derived mesenchymal stem cells (ADMSC) and ADMSC-derived exosomes markedly reduced brain infarct volume and preserved neurological function in rat after acute ischemic stroke. Oncotarget. 2016 Nov 15;7(46):74537-74556. doi: 10.18632/oncotarget.12902. PMID 27793019
- [Background] Doeppner TR, Herz J, Gorgens A, Schlechter J, Ludwig AK, Radtke S, de Miroschedji K, Horn PA, Giebel B, Hermann DM. Extracellular Vesicles Improve Post-Stroke Neuroregeneration and Prevent Postischemic Immunosuppression. Stem Cells Transl Med. 2015 Oct;4(10):1131-43. doi: 10.5966/sctm.2015-0078. Epub 2015 Sep 3. PMID 26339036
- [Background] Zhang Y, Chopp M, Liu XS, Katakowski M, Wang X, Tian X, Wu D, Zhang ZG. Exosomes Derived from Mesenchymal Stromal Cells Promote Axonal Growth of Cortical Neurons. Mol Neurobiol. 2017 May;54(4):2659-2673. doi: 10.1007/s12035-016-9851-0. Epub 2016 Mar 19. PMID 26993303
- [Background] Stonesifer C, Corey S, Ghanekar S, Diamandis Z, Acosta SA, Borlongan CV. Stem cell therapy for abrogating stroke-induced neuroinflammation and relevant secondary cell death mechanisms. Prog Neurobiol. 2017 Nov;158:94-131. doi: 10.1016/j.pneurobio.2017.07.004. Epub 2017 Jul 23. PMID 28743464
- [Background] Parekkadan B, Milwid JM. Mesenchymal stem cells as therapeutics. Annu Rev Biomed Eng. 2010 Aug 15;12:87-117. doi: 10.1146/annurev-bioeng-070909-105309. PMID 20415588
- [Background] Chen G, Luo X, Qadri MY, Berta T, Ji RR. Sex-Dependent Glial Signaling in Pathological Pain: Distinct Roles of Spinal Microglia and Astrocytes. Neurosci Bull. 2018 Feb;34(1):98-108. doi: 10.1007/s12264-017-0145-y. Epub 2017 Jun 5. PMID 28585113
- [Background] Rayasam A, Hsu M, Kijak JA, Kissel L, Hernandez G, Sandor M, Fabry Z. Immune responses in stroke: how the immune system contributes to damage and healing after stroke and how this knowledge could be translated to better cures? Immunology. 2018 Jul;154(3):363-376. doi: 10.1111/imm.12918. Epub 2018 Mar 26. PMID 29494762
- [Background] Wang Z, He D, Zeng YY, Zhu L, Yang C, Lu YJ, Huang JQ, Cheng XY, Huang XH, Tan XJ. The spleen may be an important target of stem cell therapy for stroke. J Neuroinflammation. 2019 Jan 30;16(1):20. doi: 10.1186/s12974-019-1400-0. PMID 30700305
- [Background] Ito M, Kuroda S, Sugiyama T, Maruichi K, Kawabori M, Nakayama N, Houkin K, Iwasaki Y. Transplanted bone marrow stromal cells protect neurovascular units and ameliorate brain damage in stroke-prone spontaneously hypertensive rats. Neuropathology. 2012 Oct;32(5):522-33. doi: 10.1111/j.1440-1789.2011.01291.x. Epub 2012 Jan 12. PMID 22239468
- [Background] Miyamoto M, Kuroda S, Zhao S, Magota K, Shichinohe H, Houkin K, Kuge Y, Tamaki N. Bone marrow stromal cell transplantation enhances recovery of local glucose metabolism after cerebral infarction in rats: a serial 18F-FDG PET study. J Nucl Med. 2013 Jan;54(1):145-50. doi: 10.2967/jnumed.112.109017. Epub 2012 Nov 30. PMID 23204494
- [Background] Chi L, Huang Y, Mao Y, Wu K, Zhang L, Nan G. Tail Vein Infusion of Adipose-Derived Mesenchymal Stem Cell Alleviated Inflammatory Response and Improved Blood Brain Barrier Condition by Suppressing Endoplasmic Reticulum Stress in a Middle Cerebral Artery Occlusion Rat Model. Med Sci Monit. 2018 Jun 11;24:3946-3957. doi: 10.12659/MSM.907096. PMID 29888735
- [Background] Ishibashi S, Sakaguchi M, Kuroiwa T, Yamasaki M, Kanemura Y, Shizuko I, Shimazaki T, Onodera M, Okano H, Mizusawa H. Human neural stem/progenitor cells, expanded in long-term neurosphere culture, promote functional recovery after focal ischemia in Mongolian gerbils. J Neurosci Res. 2004 Oct 15;78(2):215-23. doi: 10.1002/jnr.20246. PMID 15378509
- [Background] Iihoshi S, Honmou O, Houkin K, Hashi K, Kocsis JD. A therapeutic window for intravenous administration of autologous bone marrow after cerebral ischemia in adult rats. Brain Res. 2004 May 8;1007(1-2):1-9. doi: 10.1016/j.brainres.2003.09.084. PMID 15064130
- [Background] Mahla RS. Stem Cells Applications in Regenerative Medicine and Disease Therapeutics. Int J Cell Biol. 2016;2016:6940283. doi: 10.1155/2016/6940283. Epub 2016 Jul 19. PMID 27516776
- [Background] Wei Y, Pu Y, Pan Y, Nie X, Duan W, Liu D, Yan H, Lu Q, Zhang Z, Yang Z, Wen M, Gu W, Hou X, Ma N, Leng X, Miao Z, Liu L; Co-Investigators. Cortical Microinfarcts Associated With Worse Outcomes in Patients With Acute Ischemic Stroke Receiving Endovascular Treatment. Stroke. 2020 Sep;51(9):2742-2751. doi: 10.1161/STROKEAHA.120.030895. Epub 2020 Aug 19. PMID 32811382
- [Background] Jia B, Ren Z, Mokin M, Burgin WS, Bauer CT, Fiehler J, Mo D, Ma N, Gao F, Huo X, Luo G, Wang A, Pan Y, Song L, Sun X, Zhang X, Gui L, Song C, Peng Y, Wu J, Zhao S, Zhao J, Zhou Z, Li Y, Jing P, Yang L, Liu Y, Zhao Q, Liu Y, Peng X, Gao Q, Guo Z, Chen W, Li W, Cheng X, Xu Y, Zhang Y, Zhang G, Lu Y, Lu X, Wang D, Wang Y, Li H, Ling L, Peng G, Zhang J, Zhang K, Li S, Qi Z, Xu H, Tong X, Ma G, Liu R, Guo X, Deng Y, Leng X, Leung TW, Liebeskind DS, Wang Y, Wang Y, Miao Z; ANGEL-ACT Study Groupdagger. Current Status of Endovascular Treatment for Acute Large Vessel Occlusion in China: A Real-World Nationwide Registry. Stroke. 2021 Apr;52(4):1203-1212. doi: 10.1161/STROKEAHA.120.031869. Epub 2021 Feb 18. PMID 33596674
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Ashour W, Al-Anwar AD, Kamel AE, Aidaros MA. Predictors of early infection in cerebral ischemic stroke. J Med Life. 2016 Apr-Jun;9(2):163-9. PMID 27453748
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Background] Pires AO, Mendes-Pinheiro B, Teixeira FG, Anjo SI, Ribeiro-Samy S, Gomes ED, Serra SC, Silva NA, Manadas B, Sousa N, Salgado AJ. Unveiling the Differences of Secretome of Human Bone Marrow Mesenchymal Stem Cells, Adipose Tissue-Derived Stem Cells, and Human Umbilical Cord Perivascular Cells: A Proteomic Analysis. Stem Cells Dev. 2016 Jul 15;25(14):1073-83. doi: 10.1089/scd.2016.0048. Epub 2016 Jun 27. PMID 27226274
- [Background] Ciervo Y, Ning K, Jun X, Shaw PJ, Mead RJ. Advances, challenges and future directions for stem cell therapy in amyotrophic lateral sclerosis. Mol Neurodegener. 2017 Nov 13;12(1):85. doi: 10.1186/s13024-017-0227-3. PMID 29132389